CLINICAL TRIAL: NCT05803993
Title: TRApianto di Microbiota Intestinale in Pazienti Affetti da Sindrome Dell'Intestino IRritabile Con Stipsi: Studio Clinico Randomizzato Controllato in Singolo Centro
Brief Title: Fecal Microbiota Transplantation to Relieve Symptoms of Irritable Bowel Syndrome With Constipation
Acronym: TRAMIR-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Cammarota Giovanni, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4475
Record Dates: First submitted 2023-03-10; First posted 2023-04-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Gut microbiota; Fecal microbiota transplantation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Recruited subjects will be randomized with 1:1 ratio to receive FMT from healthy donors or autologous FMT (placebo). Patients will be evaluated before FMT and after 30, 60, 90 and 365 days
Who Masked: Participant, Investigator
Masking Description: The collected data will be analyzed in blind, as only one person not involved in the activities related to all the procedures of the study will know if faeces will be infused from a healthy donor or if an autologous FMT will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT from healthy donor (Experimental): Subjects receiving a single infusion FMT via colonoscopy from healthy donor
  Interventions: Procedure: Fecal microbiota transplantation (FMT) Single FMT infusion
- Autologous FMT (Placebo Comparator): Subjects receiving a single infusion autologous FMT via colonoscopy
  Interventions: Procedure: Fecal microbiota transplantation (FMT) Single FMT infusion

INTERVENTIONS:
Procedure: Fecal microbiota transplantation (FMT) Single FMT infusion — Single FMT infusion via colonoscopy

SUMMARY:
Irritable bowel syndrome (IBS) is a complex multifactorial functional disorder, whose pathophysiology is largely associated to an impairment of the intestinal microbiota composition, namely dysbiosis. Thus, the modulation of the gut microbiota has been proposed as a possible therapeutic strategy for IBS patients alongside with current available drugs. Fecal microbiota transplantation (FMT) is a promising strategy to restore intestinal eubiosis. In this randomised double-blind placebo-controlled trial patients diagnosed with IBS with constipation are assigned with 1:1 ratio to receive FMT from healthy donor or autologous FMT (placebo group) to assess the effectiveness of FMT on IBS symptoms and quality of life, to evaluate the safety of FMT among IBS patients and to estimate any change in the gut microbiota composition of IBS patients after the FMT.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common chronic functional disorder with a prevalence varying between 10 and 15%. IBS is characterized by recurrent chronic abdominal pain associated with altered defecation. Intestinal dysbiosis is thought to be one of the major drivers in IBS pathophysiology, since several studies have shown that there are substantial differences in microbial composition between IBS patients and healthy subjects. Moreover, the modulation of the gut microbiota in IBS patients seems a promising therapeutic approach, since a benefit on symptoms with certain antibiotics, probiotics, prebiotics, synbiotics and diet has been reported. Fecal microbiota transplantation (FMT) from healthy donors is generally considered a safe and well-tolerated procedure ant it is described to be capable of restoring eubiosis of the recipient in the long term. Recently, a certain effectiveness of FMT in ameliorating intestinal symptoms, psychological aspects and quality of life alongside with a restoration of eubiosis among IBS patients has been described. This is a prospective randomized double-blind placebo-controlled trial aimed at estimating the benefits of FMT among IBS patients with constipation. The assessment of the effectiveness on IBS symptoms and quality of life, the evaluation of the safety and the changes in the gut microbiota composition (performed with shotgun sequencing techniques) among IBS patients will be evaluated before after the FMT. 35 patients will be enrolled in 24 months. Recruited subjects will be randomized with 1:1 ratio to receive FMT from healthy donors or autologous FMT (placebo). The effectiveness of FMT in improving the IBS symptoms and IBS-related quality of life will be estimated with the IBS-SSS and IBS-QOL questionnaire, respectively, before FMT and after 30, 60, 90 and 365 days. Moreover, the frequency and form of evacuations according to the Bristol scale will be recorded at the same timepoints from diaries provided to the patients. Changes in gut microbiota composition will be estimated by comparing the composition of the faecal microbiota of the recipient before and 90 days after the FMT. The data will be evaluated using Intention-to-treat (ITT) statistical analysis and per-protocol (PP) analysis. Difference between the two groups will be calculated by two-tailed tests, Wilcoxon-Rank Sum Test for continuous variables and by the Fisher's exact probability test for categorical variables. The response rate to FMT will be evaluated by the Fisher's exact test. Adverse events will be assessed. The composition of the faecal microbiota of the recipient before and after the FMT will also be analysed and also compared with the healthy donor's one using the UniFrac method.

ELIGIBILITY:
Inclusion Criteria:

* Ability to express and give informed consent
* Age ≥ 18 years
* Diagnosis of constipation-predominant or with mixed/alternating stool pattern IBS, according to the Rome IV criteria
* Have performed a colonoscopy within the last 5 years that has ruled out intestinal diseases

Exclusion Criteria:

* Taking antibiotics or probiotics within the 8 weeks before the baseline visit
* Patients with chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis, indeterminate colitis or eosinophilic gastroenteritis), malignant neoplasms of the gastroenteric tract, celiac disease, diverticular disease
* Uncontrolled heart failure or severe heart disease with EF < 30%
* Severe respiratory failure
* Serious psychiatric conditions or psychological instability according to the clinician
* Contraindication to fecal microbiota transplantation (high risk of complications related to colonoscopy)
* Previous abdominal surgery on the gastroenteric tract (except cholecystectomy, appendectomy and other types of surgery not involving the digestive tract)
* Patients with cutaneous enterostomy
* Pregnancy or lactation
* Concurrent enrollment in other interventional experimental protocols
* Personality unstable or unable to adhere to protocol procedures
* Any clinical condition which, in the opinion of the investigators, may contraindicate enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Improving IBS symptoms assessed with the IBS severity scoring system (IBS-SSS) | 365 days
  To assess the effectiveness of healthy donor FMT in improving the symptoms of IBS without constipation compared to autologous microbiota transplantation using the IBS-SSS (< 175: mild IBS; 175-300: moderate IBS; > 300: severe IBS)
Number and severity grade of adverse events after FMT | 365 days
  To assess the number and severity grade of adverse events occurred after FMT

SECONDARY OUTCOMES:
Quality of life related to IBS evaluated with the IBS Quality of Life (IBS-QOL) questionnaire | 365 days
  To assess the effectiveness of healthy donor gut microbiota transplantation in improving the quality of life of patients with IBS without constipation compared to autologous FMT using the IBS-QOL questionnaire (range: 34-170; lower scores indicate better IBS-QoL)
Engraftment of donor microbiota after FMT, evaluated through the 16s rRNA sequencing | 365 days
  Changes in the fecal microbiota of the recipients after FMT from healthy donor or autologous microbiota transplantation will be evaluated through the 16s rRNA sequencing and compared to the baseline condition

CONTACTS AND LOCATIONS:
Locations (1):
- Giovanni Cammarota, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ianiro G, Masucci L, Quaranta G, Simonelli C, Lopetuso LR, Sanguinetti M, Gasbarrini A, Cammarota G. Randomised clinical trial: faecal microbiota transplantation by colonoscopy plus vancomycin for the treatment of severe refractory Clostridium difficile infection-single versus multiple infusions. Aliment Pharmacol Ther. 2018 Jul;48(2):152-159. doi: 10.1111/apt.14816. Epub 2018 May 30. PMID 29851107
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Ianiro G, Valerio L, Masucci L, Pecere S, Bibbo S, Quaranta G, Posteraro B, Curro D, Sanguinetti M, Gasbarrini A, Cammarota G. Predictors of failure after single faecal microbiota transplantation in patients with recurrent Clostridium difficile infection: results from a 3-year, single-centre cohort study. Clin Microbiol Infect. 2017 May;23(5):337.e1-337.e3. doi: 10.1016/j.cmi.2016.12.025. Epub 2017 Jan 3. PMID 28057560
- [Background] Cammarota G, Ianiro G, Magalini S, Gasbarrini A, Gui D. Decrease in Surgery for Clostridium difficile Infection After Starting a Program to Transplant Fecal Microbiota. Ann Intern Med. 2015 Sep 15;163(6):487-8. doi: 10.7326/L15-5139. No abstract available. PMID 26370022
- [Background] Cammarota G, Masucci L, Ianiro G, Bibbo S, Dinoi G, Costamagna G, Sanguinetti M, Gasbarrini A. Randomised clinical trial: faecal microbiota transplantation by colonoscopy vs. vancomycin for the treatment of recurrent Clostridium difficile infection. Aliment Pharmacol Ther. 2015 May;41(9):835-43. doi: 10.1111/apt.13144. Epub 2015 Mar 1. PMID 25728808